CLINICAL TRIAL: NCT01044953
Title: Repercussions of a Shortened Winter Break on Injury Incidence Within the German Professional Soccer Leagues
Brief Title: Injury Incidence in Professional Soccer
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Collaborators: Deutsche Fußball-Liga GmbH (German Soccer League Ltd.) (Unknown)
Responsible Party: Dr. med. Karen aus der Fünten, Saarland University, Institute for Sports and Preventive Medicine
Other Study IDs: sportmed-saarland-01/2009
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Injury
Keywords: injury incidence; male professional soccer; Change of injury incidence in professional soccer
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Soccer Players: German professional soccer players
  Interventions: Other: shortened winter break

INTERVENTIONS:
Other: shortened winter break — winter break shortened by 3 weeks (from 6.5 to 3.5) within the German Professional Soccer League in season 2009/2010

SUMMARY:
The winter break within the German Professional Football Leagues will be shortened as for the season 2009/2010 from 6.5 to 3.5 weeks. That might have repercussions on injury incidence in either way, positive or negative. On the one hand, recovery time during the winter will be shorter, which might lead to an increased risk of injury. On the other hand, it will allow a better spread of games in the second round, thus reducing the amount of the so-called "English weeks", which in turn could reduce the number of injuries. This study compares injury incidence between the season 2008/2009 (long winter break) and the season 2009/2010(short winter break) via questionnaires in accordance with UEFA/FIFA injury evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

* German professional male soccer players

Exclusion Criteria:

* Loss of professional status as a soccer player

Ages: 16 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: German professional male soccer players
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
injury incidence | 2 seasons

SECONDARY OUTCOMES:
types of injury | 2 seasons

CONTACTS AND LOCATIONS:
Overall Officials: Karen aus der Fünten, MD, MChiro, Principal Investigator — Saarland University, Institute for Sports and Preventive Medicine